CLINICAL TRIAL: NCT00664040
Title: Heredity and Phenotype Intervention (HAPI) Heart Study
Acronym: HAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Braxton Mitchell, PI, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00040375; U01HL072515 (NIH); U01HL072515-05 (NIH); HP-00040375 (Other: University of Maryland, Baltimore)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aspirin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Aspirin — The aspirin intervention (81 mg per day) will last a total of 14 days. Pills will be provided in a pre-loaded pillbox. The field team will visit the subject at his/her home at least once to insure adherence to the aspirin intervention and to monitor for adverse side effects. On day 14 of the aspirin intervention, the subject will visit the clinic for a fasting blood draw for platelet aggregation and inflammatory marker studies. A pill count will be performed to assess adherence. The subject can miss up to four aspirin doses over the two-week period; however, an aspirin must be taken each day for the three days prior to clinic visit 2. The aspirin intervention can be extended for up to three days (17 days total) to meet the latter criteria. If more than four doses were missed, then the physician should be contacted and the patient should be withdrawn from the aspirin intervention. Platelet aggregation will be measured 1 hour after the last dose of aspirin.
Other: Cold Pressor Test — This intervention consists of the participant placing his or her hand and wrist into ice water for 2½ minutes. The blood pressure is taken before and after the arm is removed from the water. An ultrasound machine is used to take pictures of the brachial artery in the left arm before and after the arm is removed from the water.
Other: High Fat Meal — The participants are given a high fat milk shake consisting of 83% fat. Blood samples are drawn from a catheter placed in the participant's arm prior to the test. The samples are drawn before the milk shake and at 1, 2, 3, 4, and 6 hours after the milk shake is consumed. Before and at 2, 4 and 6 hours following the meal the ultrasound is used to obtain images of the brachial artery.
Other: Dietary Salt — The salt intervention will consist of 6 days of an isocaloric high salt diet (270 mmol/d) followed by a washout period of at least 8 days and then a low salt diet (40 mmol/d). All food will be prepared by a registered dietician and dietary technicians in a specially equipped kitchen. The specific foods will consist of approximately 50% carbohydrates, 35% fat, and 15% protein. Dietary potassium will remain constant at 120 mmol/d. A food diary will be kept for each diet and subjects will be instructed to eat only the food provided. A field nurse will visit the home on days 3 and 5 of each diet to insure that neither diet is acutely affecting the health status of the subject. A first AM void spot urine will be obtained to measure sodium, potassium and creatinine on the 4th, 5th, and 6th days of each diet to insure compliance. Blood pressure will be measured using an ambulatory blood pressure monitor for 24 hours on the last day of each diet.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States and many people that die of heart disease have no previous symptoms. This study will look specifically at the response to four short-term environmental exposures including: the body's response to a cold stimulus, to a high fat milk shake, to aspirin, and to a high and low salt diet. These interventions are all known to influence CVD and people can have different responses to these interventions, which may be due, at least in part, to differences in genetic make up.

DETAILED DESCRIPTION:
Nearly one million Americans died of CVD in 1999, and it is predicted that, over one million Americans will have a myocardial infarction (MI) with 650,000 of these experiencing their first MI. Coronary artery disease (CAD) is the leading cause of mortality in the U.S., accounting for 1 of every 5 deaths, or 680,000 of more than 2,000,000 deaths. CAD is also the leading cause of premature, permanent disability in the U.S. labor force, accounting for more than $110 billion in health care costs annually, as compared to $329 billion for all CVD. Risk factors for CAD include high blood pressure, tobacco smoke, abnormal lipids and lipoproteins, physical inactivity, overweight and obesity, diabetes mellitus, increasing age, male sex, heredity, individual response to stress, and menopause in women. Other indicators for increased risk of events include the presence and extent of coronary artery calcification, endothelial dysfunction, and platelet aggregation. Of those who die suddenly from CAD, 50% of men and 63% of women have no previous symptoms. Studies of how specific environmental interventions may interact with genes to influence selected risk factors, especially in individuals with varying extent of vascular calcification, a marker of atherosclerosis, will facilitate the early identification of asymptomatic high-risk individuals who will benefit from existing or new interventions.

The overall objective of this proposal is to identify novel loci (and ultimately genes) that interact with specific environmental exposures to modify risk factors for cardiovascular disease (CVD). To achieve this goal, we will perform four short-term interventions known to modify CVD risk in participants of the Amish Family Calcification Study (AFCS), an ongoing study of the joint genetic determinants of CVD and osteoporosis. Over 1,000 individuals from this ongoing study have already been recruited and are being characterized with respect to CVD risk factors, including blood pressure, body composition, lipids, and coronary artery calcification (by electron beam computerized tomography (EBCT)). From a previous examination, DNA has been collected on all AFCS subjects and a 5-cM genome scan (~800 short tandem repeat (STR) markers) has been completed by the NHLBI Mammalian Genotyping Service. Thus, this large family study from a unique genetically homogeneous founder population provides an ideal opportunity to identify genes that interact with the environment in shaping risk factors for CVD. The Specific Aims of this proposal are:

1. To perform four focused short-term interventions known to affect cardiovascular function in 1,000 subjects from the AFCS. Responses of relevant CVD-related quantitative traits will be measured. The interventions and responses will be: a. cold pressor stress and changes in blood pressure and changes in endothelial function as assessed by brachial artery dilation (BART); b. a high fat load and changes in brachial artery flow mediated dilation (FMD) and serum lipid levels; c. high salt and low salt diets and changes in blood pressure; and d. aspirin and changes in platelet function and inflammatory markers.
2. To characterize the genetic epidemiology of the responses to each short-term intervention by: a. estimating the heritability of each response to the intervention; b. determining if response to intervention is correlated with coronary artery and aortic calcification and if so, if the association can be explained by common genes or shared environments; and c. determining if response to intervention is correlated with baseline measures of CVD risk factors, and if so, if the association can be explained by common genes or shared environments.
3. To identify specific chromosomal loci that influence CVD-related trait responses to the four short-term interventions by performing genome-wide linkage analysis utilizing a 5 cM density (~800 STR markers) genetic map already available in 1,000 subjects of the AFCS.
4. To determine if chromosomal regions linked to, or associated with, variation in CVD-related trait responses are also linked to, or associated with, variation in coronary artery or aortic calcification.
5. To fine map the putative chromosomal loci linked to variation in CVD-related trait responses to short-term environmental interventions through linkage disequilibrium mapping with closely spaced single nucleotide polymorphism (SNP) markers.

ELIGIBILITY:
Inclusion Criteria:

Participant of Amish Family Calcification Study or related to a AFCS participant and at least 20 years old.

Exclusion Criteria:

Excluded for the entire study if the subject-

1. Is currently pregnant; however they will become eligible six months after delivery.
2. Has severe hypertension (bp > 180/105), making it unethical not to recommend prompt treatment.
3. Takes medications that would affect the outcome(s) to be measured and cannot willingly and safely, in the opinion of the treating physician and study physician, discontinue these medications for 1 week prior to protocol initiation. These medications include anti-hypertensive agents (e.g., beta-blockers, calcium channel antagonists, ACE inhibitors, and diuretics), lipid lowering agents, nitrates, systemic glucocorticoids, adrenergic or cholinergic-acting agents including cold formulas and antidepressants, and diet/weight loss agents.
4. Is taking vitamins and are unwilling to discontinue their use for at least 1 week prior to study.
5. Has a coexisting malignancy
6. Has a creatinine greater than 2.0, AST or ALT greater than 2 times the upper limit of normal, Hct less than 32, or a TSH less than 0.4 or greater than 5.5.

Excluded from the Cold Pressor Test if the subject-

1. Has Raynaud's disease or symptoms

Excluded from the High Fat Challenge if the subject-

1. Has a malabsorption disorder or lactose intolerance
2. Has symptoms of gall bladder disease or history of pancreatitis

Excluded from the Dietary Salt Intervention if the subject-

1. Has stage III or greater congestive heart failure
2. Has food allergies to foods included in the diet

Excluded from the Aspirin Intervention if the subject-

1. Has a bleeding disorder or history of gastrointestinal bleeding
2. Has a blood pressure greater than 160/95
3. Is currently taking aspirin and have conditions that might place them at increased risk from aspirin withdrawal 14 days prior to protocol initiation, including history of unstable angina, MI, angioplasty (including stent placement), coronary artery bypass surgery, atrial fibrillation, stroke or transient ischemic attacks, type 2 diabetes, or deep vein thrombosis or other thrombosis
4. Has polycythemia, or thrombocytosis (platelet count greater than 500,000)
5. Has thrombocytopenia (platelet count less than 75,000)
6. Has had surgery within the last 6 months
7. Has an aspirin allergy
8. Is currently breast feeding
9. Aggregation with Collagen 5 micrograms/mL is less than 7 ohms or greater than 31 ohms, OR no aggregation at baseline with arachadonic acid

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2003-05; Study Completion 2006-08 (Actual)